CLINICAL TRIAL: NCT03115372
Title: The National Center for Reducing Asian American Cancer Health Disparities Research Project on Lay Health Workers and Asian Americans (AANCART)
Brief Title: Lay Health Worker Outreach in Increasing Colorectal Cancer Screening in Asian Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11056; NCI-2017-00515 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA153499 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Carcinoma; Health Status Unknown; Healthy Subject
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (CRC education) (Experimental): LHWs undergo training over 3 days and recruit 15 participants from their social network. Participants attend a CRC educational session conducted by an LHW over 90 minutes at month 1 and 3. Participants receive phone calls from the LHW at months 2 and 4 reminding them about CRC screening.
  Interventions: Other: Educational Intervention; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Group II (CRC brochure) (Active Comparator): LHWs undergo training over 3 days and recruit 15 participants from their social network. Participants attend a lecture on healthy nutrition for cardiovascular health presented by a professional health educator at months 1 and 3. After the first meeting, participants receive a brochure on CRC screening. Participants receive phone calls from the LHW at months 2 and 4 regarding changes in their nutritional behavior. Participants may attend an optional post-intervention LHW outreach session on CRC screening.
  Interventions: Other: Educational Intervention; Other: Informational Intervention; Other: Survey Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Educational Intervention — Attend CRC education session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (CRC education)
Other: Educational Intervention — Attend healthy nutrition session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (CRC brochure)
Other: Informational Intervention — Receive CRC screening brochure
  Arms: Group II (CRC brochure)
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive telephone reminder about CRC screening
  Arms: Group I (CRC education)
Behavioral: Telephone-Based Intervention — Receive telephone reminder about healthy nutrition
  Arms: Group II (CRC brochure)

SUMMARY:
This randomized clinical trial studies how well a lay health worker outreach works in increasing colorectal cancer screening in Asian Americans. Training community members to educate participants about colorectal cancer and its prevention may improve colorectal cancer screening rates in Asian Americans.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the efficacy of lay health worker (LHWs) outreach on colorectal cancer (CRC) screening among 3 Asian American groups (Filipinos, Hmong, and Koreans) in a cluster randomized controlled trial (RCT) comparing CRC education delivered by LHWs (intervention) to a CRC brochure and nutrition education (control).

II. Examine the processes through which LHWs communicate with, connect to, and convince community members from 3 Asian American cultures of the importance of CRC screening using mixed methods.

OUTLINE: Lay health workers (LHWs) are randomized to 1 of 2 groups.

GROUP I (CRC EDUCATION): LHWs undergo training over 3 days and recruit 15 participants from their social network. Participants attend a CRC educational session conducted by an LHW over 90 minutes at month 1 and 3. Participants receive phone calls from the LHW at months 2 and 4 reminding them about CRC screening.

GROUP II (CRC BROCHURE): LHWs undergo training over 3 days and recruit 15 participants from their social network. Participants attend a lecture on healthy nutrition for cardiovascular health presented by a professional health educator at months 1 and 3. After the first meeting, participants receive a brochure on CRC screening. Participants receive phone calls from the LHW at months 2 and 4 regarding changes in their nutritional behavior. Participants may attend an optional post-intervention LHW outreach session on CRC screening.

After completion of the study, patients are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* LHW: self-identified as Filipino, Hmong, or Korean Americans
* LHW: age 18 or older
* LHW: are fluent in a Filipino language (Tagalog or Ilocano), Hmong, Korean, or English
* LHW: Live in the relevant area and intend to stay there for the next 12 months
* PARTICIPANTS: Self-identified as Filipino, Hmong, or Korean Americans
* PARTICIPANTS: speak a language that the LHW can speak such as Tagalog, Ilocano, Hmong, Korean, or English
* PARTICIPANTS: live in relevant area and intend to stay there for at least 12 months
* PARTICIPANTS: Are willing to participate in a study about health behaviors involving nutrition or CRC screening

Exclusion Criteria:

* Personal history of CRC
* Medical problems which may prevent them from attending 2 educational sessions

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 982 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who report ever having had a CRC screening test | Baseline to 6 months
  Bivariable and multivariable analyses of the binary outcomes (CRC screening ever, up-to-date, and intention) will be conducted using generalized linear models to evaluate the efficacy of the intervention. A linear model with identity link function will be used with group (intervention or control), time (pre- or post-), and group-by-time interaction to test for a difference in the change from pre- to post-intervention between the 2 groups, thus measuring the efficacy of the intervention.

SECONDARY OUTCOMES:
Proportion of participants who are up-to-date for CRC screening | At 6 months
  Bivariable and multivariable analyses of the binary outcomes (CRC screening ever, up-to-date, and intention) will be conducted using generalized linear models to evaluate the efficacy of the intervention.
Proportion of participants who intend to obtain CRC screening in the next 6 months | At 6 months
  Bivariable and multivariable analyses of the binary outcomes (CRC screening ever, up-to-date, and intention) will be conducted using generalized linear models to evaluate the efficacy of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tung Nguyen, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Hawaii Cancer Center, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: No